CLINICAL TRIAL: NCT03140098
Title: Evaluation of the Tolerance and Efficacy of COVA™+ CARD in Adult Cardiac Surgery. A Prospective, Observational and Single Center Study.
Brief Title: Evaluation of COVA™+ CARD in Adult Cardiac Surgery
Status: Withdrawn | Type: Observational
Why Stopped: Decision not to pursue
Sponsor: Biom'Up France SAS (Industry)
Responsible Party: Sponsor
Other Study IDs: ETC 2017-002
Record Dates: First submitted 2017-04-26; First posted 2017-05-04 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Safety; Tolerance
Keywords: Collagen membrane; Cardiac surgery; Postoperative complication
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: cardiac surgery requiring a collagen membrane COVA™+ — At the end of the cardiac surgery, the collagen membrane is implanted on the dissection area in order to prevent the formation of postoperative adhesions.

SUMMARY:
The aim of this observational study is to evaluate the safety of the guided healing and adhesion prevention membrane, COVA™+ CARD, in adult cardiac surgery. The causality of the collagen membrane according to the occurrence of peri and post-operative complications will be evaluated.

DETAILED DESCRIPTION:
Assessment of the safety of COVA™+ CARD, collagen membrane to prevent adhesion appearance, in cardiac surgery in adult patients:

* collection of post-operative complications, causality of the membrane
* collection of complications in the 3-month period after the surgery, causality of the membrane
* collection of peri-operative complications, causality of the membrane
* collection of complications, 3 months after the surgery
* assessment of the efficacy of COVA™+ CARD if re-operation
* assessment of the surgeon's satisfaction

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Cardiac surgery using COVA™+ CARD

Exclusion Criteria:

* In accordance with the instruction for use (IFU) of the medical device.
* Refusal of participation to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who will undergo a cardiac surgery.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-02 (Estimated); Primary Completion 2018-02 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the tolerance of COVA™+ CARD in cardiac surgery | 3 months
  Recording of complications reported in the 3-month postoperative period and determination of the causality of the collagen membrane.

SECONDARY OUTCOMES:
Evaluation of the tolerance of COVA™+ CARD in cardiac surgery | Hospitalization stay (up to 30 days)
  Recording of the immediate postoperative complications and determination of the causality of the collagen membrane.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Madonna, Principal Investigator — University Hospital, Bordeaux

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Potential interest of a new absorbable collagen membrane in the prevention of adhesions in paediatric cardiac surgery — https://www.ncbi.nlm.nih.gov/pubmed/23906681